CLINICAL TRIAL: NCT04080362
Title: A Prospective, Multicenter, Single Group Assignment Study for Evaluating the Safety and Effectiveness of MitralStitch Mitral Valve Repair System in Patients With Moderate to Severe and Severe Mitral Regurgitation.
Brief Title: Safety and Performance Study of the MitralStitch Repair System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRACLE_II
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-05

CONDITIONS: Mitral Regurgitation
Keywords: Mitral Regurgitation; Mitral Valve Repair; Transapical
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: The clinical trial was designed as a single group assignment study. The participants with moderate to severe and severe mitral valve regurgitation will receive a transapical beating-heart mitral valve repair surgery using MitralStitchTM mitral valve repair system.
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MitralStitch repair system (Experimental): Experimental group is allocated to use novel mitral vavle repair system manufactured by Hangzhou Valgen Medtech Co., Ltd
  Interventions: Device: MitralStitch

INTERVENTIONS:
Device: MitralStitch — With transesophageal echocardiographic guidance,implanting ePTFE sutures as artificial neochordae or ege-to-ege repair using MitralStitch System

SUMMARY:
The main objective is to assess the effectiveness and safety of the MitralStitch repair system in patients with moderate to severe and severe mitral regurgitation.

DETAILED DESCRIPTION:
The clinical trial was designed as a prospective, multicenter, single group assignment study. The participants with moderate to severe and severe mitral valve regurgitation will receive a transapical beating-heart mitral valve repair surgery using MitralStitch mitral valve repair system after signed the informed consent. The follow-up will be conducted after 30 days, 3 months, 6 months and 12 months of the operation.

The following conditions evaluate the performance of the system and the safety and efficiency of using MitralStitch mitral valve repair system in treating patients with severe mitral regurgitation.

The none occurrence of these conditions will be approved as the main validity index: death, mitral valve related surgery without mitral valve failure and moderate or severe mitral regurgitation (MR > 2+). The secondary validity index was technical success rate, instrument success rate, surgical success rate, cardiac function improvement and quality of life improvement. And the safety evaluation indicators were assessed by the incidence of major adverse events, adverse events, serious adverse events, and device defects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 yrs
2. Moderate to severe (3+) or severe (4+) mitral valve regurgitation confirmed by echocardiography (defined as MR >2+);
3. NYHA functional class II-V (Appendix 3);
4. Anatomically suitable for mitral valve repair;
5. 40mm ≤LVESD≤55 mm; 25% ≤LVEF ≤60%; tolerable for small incision thoracic surgery;
6. Mitral valve diameter ≤45mm;
7. The independent expert committee of this study determined that surgical operation was contraindicated or high-risk, and the recommended reference standard was: surgical valve replacement with STS score ≥ 8； or surgical valve repair with STS score ≥ 6； or other risk factors (e.g., There are at least two moderate to severe indicators of weakness; potential operational disorders; at least major organ dysfunction that cannot be improved after surgery, etc.)
8. The subject or the subject's legal representative fully understand and agree to join to the clinic trial.

Exclusion Criteria:

1. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
2. Severe mitral valve calcification;
3. Concomitant with greater than moderate aortic stenosis or regurgitation;
4. Mitral regurgitation caused by special pathological mechanisms, such as leaflet perforation and leaflet fissure;
5. Severe untreated coronary artery stenosis requiring revascularization; or with other cardiovascular disease requiring surgical treatment;
6. Hypertrophic cardiomyopathy with or without obstruction, restrictive cardiomyopathy, constrictive pericarditis, or other structural heart diseases that cause heart failure in patients expect dilated cardiomyopathy;
7. Myocardial infarction was performed within 4 weeks before the intervention;
8. Any vascular intervention, cardiac surgery, cardiac resynchronization therapy (CRT, CRT-D), and an implantation of implantable cardioverter defibrillator (ICD) were performed within 30 days before the intervention;
9. Any heart transplantation, mitral valve surgery or percutaneous mitral valve operation were performed before the intervention;
10. Life expectancy is less than 12 months;
11. History of, or active, rheumatic heart disease;
12. Active phase of bacterial endocarditis;
13. The active infections require concurrent antibiotic treatment;
14. History of acute peptic ulcer or upper gastrointestinal bleeding within 3 months;
15. Dysplasia of the blood system, including granulocytopenia (WBC < 3×109/L), acute anemia (HB < 90g/L), thrombocytopenia (PLT < 50×109/L), hemorrhagic constitution, and coagulopathy；
16. Modified Rankin scale ≥4；
17. Pregnant or lactating women;
18. The subject is suffered from a disease which may cause difficulty in evaluating the treatment (e.g., cancer, infection, severe metabolic disease, psychosis, etc.); or special cases were evaluated by the local experimental center heart team as not suitable for the surgical application of this clinical trial instrument;
19. Participants who have participated in clinical trials of any drug and/or medical device within 1 month before this study;
20. In the judgment of the Investigator, patients were not compliant enough to complete the study as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The success rate | 1 year
  Combined incidence of freedom from: death, surgery for Valve Dysfunction, and MR > 2+ (moderate to severe (3+) or severe (4+) mitral regurgitation) at 12 months

SECONDARY OUTCOMES:
The instant procedural success | Immediately after repair
  Technical success is defined as the absence of death, the successful implantation of the device and complete retraction of the delivery system without any need for emergency surgery or secondary intervention (including device related and surgical approach related
The success of the repair system | 12 months
  The success rate of the device is defined as the successful delivery and implantation of the device, and the successful withdrawal of the implanted parts after the completion of the release, without any technical failure or complications related to the device.
The success of the surgery | 1 month
  Surgical success was defined as the success of the instrument, MR 2+, and no major adverse events related to the instrument or operation occurred during the follow-up period after the implantation of the instrument.
New York Heart Association (NYHA) class | 12 months
  NYHA grading was used to evaluate the cardiac function status of subjects
Living quality | 12 months
  Postoperative SF-12 was used to evaluate the quality of life of the subjects
Incidence of major adverse events(MAE) | 12 months
  MAE definition: Any complications related to devices or surgeries, including but not limited to: death, emergency surgery, severe cardiac tamponade requiring pericardiocentesis or operation, hemorrhage, stroke related to operation.

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, Principal Investigator — Chinese Academy of Medical Science, Fuwai Hospital
Locations (1):
- Structural Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality, China